CLINICAL TRIAL: NCT01213394
Title: A 6-month, Prospective, Open-label, Randomized, Controlled, Pilot Study Evaluating the Efficacy, Safety and Toxicity of an Optimized Immunosuppressive Regimen of CellCept (Mycophenolate Mofetil, MMF) and Reduced Doses of Both Calcineurin-inhibitors and Prednisone in Renal Transplant Recipients With an Increased 10-year Coronary Heart Disease Risk
Brief Title: Mycophenolate Mofetil for Reducing Cardiovascular Risk in Renal Transplant Recipients
Acronym: MMCR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment.
Sponsor: Ramesh Prasad (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor-Investigator, Ramesh Prasad, Staff Nephrologist, Unity Health Toronto
Organization: Unity Health Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ML25073
Record Dates: First submitted 2010-09-28; First posted 2010-10-04 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Kidney Transplantation; Cardiovascular Diseases
Keywords: Framingham score; kidney transplant; immunosuppression; cardiovascular disease; CellCept; mycophenolate mofetil
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CellCept optimization (Experimental)
  Interventions: Drug: mycophenolate mofetil
- Control (Active Comparator)
  Interventions: Other: standard immunosuppression

INTERVENTIONS:
Drug: mycophenolate mofetil — Introduction of CellCept or increase in the dose of CellCept to a maximum of 2 g/day. In patients not already receiving CellCept, azathioprine (AZA), enteric-coated mycophenolate sodium (EC-MPS) or sirolimus (SRL) will be discontinued and replaced by CellCept in divided doses to a maximum of 2 g/day. CNI doses will be reduced to conform to the target trough levels in the low-dose CNI arms of the ELITE-Symphony study +/- steroid dose reduction. Any CNI dose change will require measurement of CNI trough levels at 7 days post dose change +/- 3 days.
  Target CNI trough levels in the Symphony study:
  * Low-dose CsA: Initial oral dose of 1-2 mg/kg bid, to achieve a target trough level of 50-100 ng/mL.
  * Low-dose TAC: Initial oral dose of 0.1 mg/kg/day divided into two doses* with a target trough level of 3-7 ng/mL (*Advagraf may also be used at a dose of 0.1 mg/kg once daily with a target trough level of 3-7 ng/mL)
  Other Names: CellCept, MMF
  Arms: CellCept optimization
Other: standard immunosuppression — Current immunosuppressive therapy will be maintained throughout the study unless a change is required for safety reasons.
  Arms: Control

SUMMARY:
The purpose of this research study is to determine if adding or increasing the dose of CellCept while lowering the dose of tacrolimus (Prograf or Advagraf) or cyclosporine (Neoral), and/or steroids can reduce the likelihood of developing coronary heart disease in the next 10 years.

The investigators will calculate the change in risk of developing coronary heart disease using the Framingham score. The Framingham score is a mathematical equation that includes the following information: Age, Gender, Diabetes status, Smoking status, Lipids, Blood Pressure. The Framingham score estimates how likely it is that someone will develop coronary heart disease over the next 10 years.

DETAILED DESCRIPTION:
Kidney transplant recipients are required to take medications called immunosuppressants to lower their immune systems to help protect the donated kidney. The medications have improved over the years and as a result the donated kidneys are generally working longer. This allows the Transplant Team to focus more on the long term complications of kidney transplantation such as cardiovascular disease.

There have been few prospective (looking forward) research studies looking at kidney transplant recipient cardiovascular risk factors after transplant.

We know that immunosuppressive medications have a number of serious side effects that can increase cardiovascular disease risk factors such as high blood pressure, high lipids (fats in the blood), and high blood sugar. Medications such as tacrolimus, cyclosporine and prednisone work well to protect the donated kidney but are also known to increase the risk of developing or worsening cardiovascular disease.

CellCept is another type of immunosuppressive agent. CellCept is not associated as much with the risk of developing cardiovascular disease.

This is a pilot study being done to collect information about cardiovascular risk factors in kidney transplant recipients and to see if adjusting the immunosuppressive medications can help to lower the overall risk for developing heart disease in the future.

This research study plans to enroll 45 participants from 2 different transplant centres in Canada: St. Michael's Hospital in Toronto and St. Paul's Hospital in Saskatoon. The study duration is approximately 7 months per participant. The study will be looking for participants who are 30 years of age or older and who are at least 6 months after the transplant operation.

ELIGIBILITY:
Inclusion Criteria:

1. Renal transplant recipients who are ≥ 6 months post-day of transplant surgery.
2. Single organ kidney recipient (may be for first or repeat transplant).
3. Age ≥ 30 years of age as of the Day 0 visit.
4. Immunosuppressive regimen consisting of a CNI (cyclosporine [CsA, Neoral] or tacrolimus [TAC, Prograf or Advagraf], corticosteroids and either MMF (CellCept), EC-MPS (Myfortic), AZA (Imuran) or SRL (Rapamune) at the baseline visit. Patients are to be maintained on the same dose(s) for at least 4 weeks prior to study enrolment.
5. If the patient is taking an MPA immunosuppressant at the time of the screening visit, the MMF (CellCept) dose must be ≤ 1500 mg/day; or the EC-MPS (Myfortic) dose must be ≤ 1080 mg/day.
6. Framingham risk factor score that exceeds the low comparative 10-year CHD risk, based on age and gender.
7. Presence of at least one established CV risk factor at baseline warranting modification of the immunosuppressive regimen including:

   * Hypertension: Blood pressure ≥ 140 mmHg systolic and/or ≥ 90 mmHg diastolic and/or requiring ≥ 1 antihypertensive medication.
   * Diabetes mellitus: Established diabetes requiring treatment with oral hypoglycemic agents or insulin, or known IFG or IGT based on 75-g oral glucose tolerance testing (2003 Canadian Diabetes Association criteria).
   * Hyperlipidemia: TC ≥ 5.2 mmol/L, or LDL-C ≥ 2.6 mmol/L, or TG ≥ 1.7 mmol/L, or TC:HDL ≥ 4 and/or requiring ≥ 1 anti-hyperlipidemia agent.
8. Willingness and ability to complete protocol requirements.
9. Written informed consent.

Exclusion Criteria:

1. Contraindication to receiving MMF (CellCept) or increasing CellCept dose.
2. Clinically suspected acute rejection (AR) or BPAR within 3 months prior to the baseline visit.
3. Proteinuria ≥ 1 g/24 hours
4. Treatment with AZA (Imuran), EC-MPS (Myfortic) or SRL (Rapamune) and patient or physician decision not to discontinue these agents and switch to MMF (CellCept) at the time of randomization.
5. MDRD (4-variable) eGFR < 15 mL/min/1.73 m2
6. Patients who currently exceed thresholds for plasma glucose, cholesterol or blood pressure. Patients may be re-considered 1 month after the treatment is in place and no further therapeutic changes are anticipated.
7. Patients who require changes to their blood pressure, blood sugar or blood lipid management between the Screening Visit and Day 0. Patients may be re-considered 1 month after the adjusted treatment is in place and no further therapeutic changes are anticipated.
8. Pregnancy, lactation or (for women of childbearing potential) inability or decision not to use a reliable method of contraception for the entire study duration.
9. Active infection requiring treatment.
10. Treatment with unlicensed investigational drugs, devices or other prohibited medications - see Section 4.4.1
11. Participation in any other interventional clinical trial during the previous 4 weeks or during this trial.
12. History of malignancy, other than non-melanoma skin cancer that has been totally excised and has not recurred for >2 years.
13. History of psychological illness or condition that could interfere with the patient's ability to understand or comply with the study requirements.
14. Presence of other significant diseases or issues which, in the opinion of the sponsor-investigator, may:

    * Put the patient at risk as a result of study participation
    * Influence the study result
    * Affect the patient's ability to participate in the study
    * Require a change in immunosuppression medication used or a dose change within the next 6 months (unstable renal function, gout that may require treatment with prednisone, etc)
    * Reduce life expectancy. Examples include but are not limited to history of noncompliance and transportation issues that could affect a participant's ability to successfully complete the study requirements. Inability or refusal to provide blood samples, end-stage disease of organs such as lung, liver or heart.
15. Exclusion of patients who are hypersensitive to CellCept (mycophenolate mofetil), mycophenolic acid or any component of the drug).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The change in the Framingham 10-yr age and gender adjusted score for coronary heart disease from baseline to Month 6 | Baseline to Month 6
The incidence of a composite of acute rejection (clinically suspected and biopsy-proven), graft loss or patient death. | Month 6

SECONDARY OUTCOMES:
Framingham point total | Baseline to Month 6
  Change in Framingham point total from baseline to month 6
Day and night blood pressure | Baseline to Month 6
  Change in day and night blood pressure (defined by awake and sleep times) measured by 24-hour ambulatory blood pressure monitoring (ABPM) from baseline to month 6
Glucose metabolism | Baseline to Month 6
  Change in glucose metabolism, based on HbA1C levels in patients with and without diabetes, and the prevalence of impaired fasting glucose (IFG) and impaired glucose intolerance (IGT) in patients without overt diabetes from baseline/randomization to month 6.
Lipid metabolism | Baseline to Month 6
  Change in lipid metabolism, measured by the fasting levels of total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) and triglycerides (TG)and ratio of TC to HDL-C from baseline/randomization to month 6
Change in renal function | Baseline to Month 6
  Change in renal function from baseline/randomization to month 6 as measured by serum creatinine, estimated glomerular filtration rate, (MDRD 4-variable equation), change in eGFR slope, change in chronic kidney disease (CKD), 24-hr urine creatinine clearance and protein/albumin excretion
Adverse cardiovascular events | Month 6
  Proportion of patients who experience any adverse cardiovascular event such as myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG), fatal and non-fatal cerebrovascular events (including fatal or non-fatal stroke, transient ischemic attack, reversible ischemic neurological deficit and subarachnoid hemorrhage). Cardiovascular events will be adjudicated by a cardiologist blinded to treatment assignment.
Highly-sensitive C-reactive protein (CRP) level | Randomization to Month 6
  Change in highly-sensitive CRP level between randomization and month 6.
Change in other biomarkers of cardiovascular risk | Randomization to Month 6
  Change in other biomarkers of cardiovascular risk between randomization and month 6: human adiponectin (including its high molecular weight isoform), uric acid, early morning urine albumin-to-creatinine ratio, B-type (brain) natriuretic peptide (BNP), fibrinogen, D-dimer (fibrin degradation fragment), advanced glycosylation endproduct (AGE), paraoxonase B, cystatin C, insulin, proinsulin, malondialdehyde (MDA), protein carbonyl, glutathione reductase/total and apolipoprotein A1, B and Lp(a).
Incidence of MMF-attributable adverse events | Month 6
  Incidence of MMF-attributable adverse events including gastrointestinal toxicities, thrombocytopenia, leucopenia and anemia.
Additional treatment with cardiovascular co-interventions | Month 6
  Requirements for additional treatment with cardiovascular co-interventions - as per guideline documents.
Opportunistic infections | Month 6
  Incidence of opportunistic infections
Malignancies | Month 6
  Incidence of malignancies
Adverse events | Month 6
  All adverse events (AEs), including clinically significant abnormalities of clinical and laboratory parameters will be captured. Summary statistics will be created for all adverse events and will be summarized by treatment group, by relation to study treatment and seriousness of the event.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ramesh Prasad, MBBS MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada